CLINICAL TRIAL: NCT06204627
Title: Effects of Transcranial Stimulation by Direct Current Associated With Laterality Trainnning in Patients With Chronic Neck Pain
Brief Title: TDCS* and Laterality Trainnning in Patients With Chronic Neck Pain
Acronym: TDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Clarice Tanaka, Director, Principal investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 94350518.6.0000.0068
Record Dates: First submitted 2020-08-27; First posted 2024-01-12 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Neck Pain; Chronic Pain
Keywords: chronic pain; neck pain; functional laterality; transcranial direct current stimulation
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The study will be controlled, randomized, double-blind and will include patients with chronic neck pain, divided into four groups:
  1. active TDCS associated with laterality recognition stimuli (n = 25);
  2. active TDCS associated with landscape recognition stimuli (n = 25);
  3. TDCS sham associated with laterality recognition stimuli (n = 25);
  4. TDCS sham associated with landscape recognition stimuli (n = 25).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be controlled, randomized and double-blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active bipolar TDCS associated with laterality recognition stimuli (Active Comparator): Participants will have carbon electrodes positioned, with contact through a 5x7cm sponge moistened in saline solution, with the anode on M1 and the cathode in the supra-orbital region. Individuals with active bipolar TDCS will receive a 2mA stimulus for twenty minutes. Meanwhile, they will use the Regognise hand application to discriminate right/left side of hand images.
  Interventions: Device: TDCS; Device: Recognize (hand) - Laterality
- Active bipolar TDCS associated with landscape recognition stimuli (Active Comparator): Participants will have carbon electrodes positioned, with contact through a 5x7cm sponge moistened in saline solution, with the anode on M1 and the cathode in the supra-orbital region. Individuals with active bipolar TDCS will receive a 2mA stimulus for twenty minutes.
  At the same time, they will be guided to recognize landscapes that do not refer to the recognition of laterality.
  Interventions: Device: TDCS; Other: Landscape recognition
- Sham TDCS associated with laterality recognition stimuli (Active Comparator): Participants will have carbon electrodes positioned, with contact through a 5x7cm sponge moistened in saline solution, with the anode on M1 and the cathode in the supra-orbital region. Stimulation will remain inactive for the 20 minutes. Meanwhile, they will use the Regognise hand app to discriminate right/left hand images.
  Interventions: Device: Recognize (hand) - Laterality; Other: Sham TDCS
- Sham TDCS associated with landscape recognition stimuli (Placebo Comparator): Participants will have carbon electrodes positioned, with contact through a 5x7cm sponge moistened in saline solution, with the anode on M1 and the cathode in the supra-orbital region. Stimulation will remain inactive for the 20 minutes. At the same time, they will be guided to recognize landscapes that do not refer to the recognition of laterality.
  Interventions: Other: Sham TDCS; Other: Landscape recognition

INTERVENTIONS:
Device: TDCS — Technique of non-invasive brain stimulation by direct current (TDCS) which involves the modulation of excitability and brain activity, capable of promoting reorganization of the cortical representation of the body schema or motor planning, and consequently, pain relief.
  Arms: Active bipolar TDCS associated with landscape recognition stimuli; Active bipolar TDCS associated with laterality recognition stimuli
Device: Recognize (hand) - Laterality — This technique stimulates the ability to recognize hand images as right/left quicklPatients with chronic pain present delayed recognition of hand laterality, which is related to the duration of symptoms and the pain evoked by the execution of the movement. Thus, this technique can have beneficial effects in breaking the pain.
  Arms: Active bipolar TDCS associated with laterality recognition stimuli; Sham TDCS associated with laterality recognition stimuli
Other: Sham TDCS — TDCS sham: The device remains inactive for 20 minutes.
  Arms: Sham TDCS associated with landscape recognition stimuli; Sham TDCS associated with laterality recognition stimuli
Other: Landscape recognition — Image recognition training that does not refer to right/left discrimination.
  Arms: Active bipolar TDCS associated with landscape recognition stimuli; Sham TDCS associated with landscape recognition stimuli

SUMMARY:
Chronic neck pain leads to decreased quality of life and absenteeism at work, generating great personal and socio-economic impact. It has been shown that patients with chronic pain have late recognition of the laterality of the hand, which is related to the duration of symptoms and pain evoked by the execution of the movement. These findings suggest that chronic pain and the consequent disuse of certain motor functions may involve a reorganization of the cortical representation of the body scheme or motor planning.

Non-invasive neuromodulation, such as transcranial direct current stimulation (TDCS), allows modulating cortical excitability and promoting pain relief.

This study intends to verify the effects of the association of noninvasive brain stimulation with TDCS with an intervention with visual and motor stimuli related to laterality in patients with neck pain.

DETAILED DESCRIPTION:
The study will be controlled, randomized, double-blind and will include patients with chronic neck pain, divided into four groups:

1. active TDCS associated with laterality recognition stimuli (n = 25);
2. active TDCS associated with landscape recognition stimuli (n = 25);
3. TDCS sham associated with laterality recognition stimuli (n = 25);
4. TDCS sham associated with landscape recognition stimuli (n = 25);

Eight induction sessions will be held twice a week for four weeks. Patients who present a positive response in the first reassessment (responders) will remain in the study follow-up and will undergo a weekly maintenance session, for four weeks, and two more biweekly sessions.

The following instruments will be used for evaluation: motor safety thresholds through a MagVenture pulse generator with a flat surface coil, figure 8; OPAL, device with sensors; Recognize™ application; Visual Analog Scale (VAS); Brief Pain Inventory (BDI); Clinical Global Impression - ICG (patient and evaluated version); Pain McGill Standard Questionnaire - Short Format; Hospital Anxiety and Depression Scale (HAD); 36-item summary health survey from the Medical Outcomes Study (SF-36); Mini best test; neurodynamic tests (upper limb tension tests); and quantitative sensory tests. In addition to the pre- and post-intervention assessments, there will be post-treatment follow-up performed three, six and 12 months after randomization by telephone or e-mail. It is expected that the combined application of tDCS with stimuli related to laterality will have positive effects in patients with neck pain, impacting on variables such as pain, functional movements and quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

* participants over 18 years old;
* pain in the cervical region, lasting more than three months and with intensity greater than 40/100 on the visual analog scale

Exclusion Criteria:

* history of seizures or epilepsy,
* history of head trauma,
* intracranial hypertension,
* intracranial metal clip,
* pregnant or breastfeeding women,
* skin lesions at the current application site;
* changes in sensitivity and allergy in the electrode positioning region.
* intermittent pain;
* Cancer;
* cardiac pacemaker;
* severe spinal diseases, such as recent fractures or ankylosing spondylitis;
* serious cardiorespiratory diseases;
* participants who refuse to sign the Free and Informed Consent Form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain symptoms | up to 3 months
  Change from Baseline in pain symptoms on the Visual Scale after treatment

SECONDARY OUTCOMES:
Clinical Global Impression | up to 3 months
  Change from Baseline in pain severity on the Clinical Global Impression scale after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No